CLINICAL TRIAL: NCT05324787
Title: Single Arm, Multi-center Clinical Trial for the Safety and Effectiveness of Venous Stent System in the Treatment of Vein Stenosis or Occlusion
Brief Title: Treatment of Vein Stenosis or Occlusion With the Oblique Stent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Endonom Medtech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GR001
Record Dates: First submitted 2022-03-31; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Iliac Vein Stenosis; Iliac Vein Occlusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Grency venous stent system (Experimental)
  Interventions: Device: Grency venous stent system

INTERVENTIONS:
Device: Grency venous stent system — Venous stent implantation during the index procedure

SUMMARY:
To evaluate the safety and effectiveness of Grency venous stent system in the treatment of iliac vein stenosis or occlusion.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the safety and effectiveness of a new dedicated venous stent system (Grency) in the treatment of iliac vein stenosis or occlusion. The Grency stent system has a hybrid oblique self-expanding design, which allows precise positioning at the iliocaval confluence.

ELIGIBILITY:
Inclusion Criteria:

1. subjects aged 18-80 years;
2. CEAP clinical grade C >=3;
3. iliac vein stenosis >=50% or occlusion;
4. patients voluntarily sign informed consent and complete follow-up.

Exclusion Criteria:

1. subjects in pregnancy or lactation;
2. renal insufficiency;
3. subjects are allergic to contrast agents and anesthetics;
4. subjects are allergic to nitinol;
5. the life expectancy of cancer patients is less than 1 year;
6. the length of the stent is expected to exceed the length of the inguinal ligament; 7. both sides of iliac vein stents were required;

8. long term bedridden or wheelchair patients; 9. the target vessel of the subject has been implanted into the iliac vein stent; 10. subjects have anticoagulant contraindications or are unable to receive long-term new oral anticoagulant therapy; 11. the investigator judged that the subjects had poor compliance and could not complete the clinical trial; 12. subjects are participating in clinical trials of other drugs or medical devices and have not yet completed the primary end point of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Patency rate of venous stent | 12 months post-intervention
  Freedom from target vessel revascularization ; freedom from in-stent stenosis more than 50% by venography.

SECONDARY OUTCOMES:
The rate of procedural technical success | During procedure
  Procedure technical success is defined as successful deployment of stent(s) to intended target without stent fracture or migration, as assessed by the investigator during the procedure.
Change in the clinical symptoms | Baseline, 3 months,6 months, and12 months post-intervention
  Change from baseline in the Venous Clinical Severity Score (VCSS) and Clinical-Etiologic-Anatomic-Pathophysiologic (CEAP) Classification at 3 months,6 months, and 12 months.
  VCSS measures 10 clinical attributes of venous disease (Pain, Varicose Veins,Venous Edema, Skin Pigmentation, Inflammation, Induration, No. Active Ulcers, Active Ulcer Size, Ulcer Duration and Compression Therapy) on a scale of 0 - 3 (Absent 0, Mild 1, Moderate 2, and Severe 3).
  Clinical-Etiologic-Anatomic-Pathophysiologic (CEAP) Classification is a system that describes a doctor's physical exam findings for vein problem(s), the cause of the problem(s), the location in the leg, and the mechanism responsible for the manifestation of the vein problem. For Clinicalclassification, the clinical components indicates disease severity, ranging from none (0 points) to active ulcers (6 points).
The rate of device related major adverse events(MAE) | 3,6,12 months post-intervention
The rate of adverse events (AE) | 3,6,12 months post-intervention

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Chinese People's Liberation Army General Hospital, Beijing
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No